CLINICAL TRIAL: NCT04741763
Title: "Night Vision and Carotenoids" A 2 Center Study of the Physiological Function of the Eyes
Brief Title: "Night Vision and Carotenoids"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Davis (Other)
Collaborators: Davis EyeCare (Other)
Responsible Party: Sponsor-Investigator, Robert Davis, co-investigator, Davis EyeCare
Organization: Davis EyeCare (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1052607-1
Record Dates: First submitted 2021-01-13; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Macular Degeneration
Keywords: Macular Disease
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Capsule type that results in null or increased MPOD (macular pigment optical density in du -density units) - either Maltodextrin Placebo or OTC commercial "Night Vision Formulation" consisting of 21 mg carotenoid capsule (14 mg zeaxanthin and 7mg lutein) supplied by www.zeavision.com (Chesterfield, MO) in research coded bottles with code held by the company. Gel caps will be supplied in a single 180 count bottle. 1 gel cap per day will be taken with a meal. Subjects will be called by telephone to improve compliance. Supplement compliance will ultimately be gauged by the number of tablets returned.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Research coded bottles with code held by the sponsor. Gel caps will be supplied in a single 180 count bottle. 1 gel cap per day will be taken with a meal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin Placebo: Experimental is 1:2
  Interventions: Dietary Supplement: EyePromise Visual Edge
- Active (Experimental): Eye Promise Visual Edge containing 8 mg zeaxanthin & 4 mg lutein Placebo: Experimental is 1:2
  Interventions: Dietary Supplement: EyePromise Visual Edge

INTERVENTIONS:
Dietary Supplement: EyePromise Visual Edge — A dietary eye supplement containing 8 mg zeaxanthin and 4 mg lutein and additional proprietary nutrients

SUMMARY:
Vision at twilight and night is more difficult and dangerous for the entire population, even more so for the elderly and especially for the elderly with degenerative disease. Multiple worldwide laboratories have demonstrated the ability to raise macular pigment optical density with dietary carotenoids. This proposal further evaluates the relationship between macular re- pigmentation and vision under stressed conditions simulating twilight and night driving.

DETAILED DESCRIPTION:
This is a study of the physiological function of the eyes at night. However, the risk of automobile injury or fatality (driver, passenger or pedestrian) associated with motor vehicle accidents has been determined to increase with age, as a result of the complex interplay of age-related declines in vision, motor and cognitive functioning. However, basic visual function is the foundation for higher order processing whether it is visual spatial or cognitive. Four recent studies reflect the cost of poor vision on driving. (www.visionimpactinstitute.org). For example, visual impairment among European drivers was examined in 2422 drivers from 5 European countries. Visual acuity, visual field, contrast sensitivity, glare sensitivity, and useful field of view were tested. Visual functions not included in the current licensing standards were found to be more impaired among drivers (compared to those functions legally required). Elderly drivers are particularly vulnerable to sensory visual impairment when driving at night, as they suffer declines in both Contrast sensitivity (CS), Glare Disability (GD) and Glare Recovery (GR).6

Justification for study involving humans

Carotenoid science is well developed with respect to the safe utilization of dietary lutein (L) /zeaxanthin (Zx) as studied by the National Institute of Health (NEI). The recently published NEI AREDS2 study- May 2013, further substantiated the safety and usefulness of prescribing the carotenoids (10 mg L / 2 mg Zx) in patients at high risk of AMD. 7 Significantly, the average American and veteran population are typically low dose consumer of these carotenoids (1 to 2 mg/day for the average American).

ELIGIBILITY:
Inclusion Criteria:

* No significant supplementary carotenoids within last 10 weeks. Without significant media opacity, cataract or congenital / acquired retinal disease other than atrophic AMD or diabetic retinopathy. Minimum 20/25 to enroll.

Exclusion Criteria:

* Unwilling or medically / psychiatrically unable to take part in a 6 month study.
* Recent ophthalmologic surgery or treatment.
* Tricare, Retirees & Enlisted Navy Personnel excluded. Already taking an OTC product to improve their night vision (containing carotenoids, polyphenols like bilberry).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
MPOD | 24 weeks
  1 degree macular pigment optic density

SECONDARY OUTCOMES:
Vimetrics Central Vision Analyzer (CVA) | 24 weeks
  measure of contrast & glare
LuxIQ- preferred luminance | 24 weeks
  preferred luminance
Useful Field of Vision (UFOV) Brain HQ | 24 weeks
  eye-brain test of functional vision and vision attention

CONTACTS AND LOCATIONS:
Overall Officials: Steven Novil, PhD, ND, Study Director — Optometry Research Lab manager, Optometry Clinic- Captain James A Lovell FHCC
Locations (2):
- United States (2):
  - The Captain James A. Lovell Federal Health Care Center (FHCC), North Chicago, Illinois
  - Davis EyeCare, Oak Lawn, Illinois